CLINICAL TRIAL: NCT03794310
Title: A Phase III Comparison Study of NPF-08 in Patients Who Receive Colonoscopy
Brief Title: Study of NPF-08 in Patients Who Receive Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NPF-08-01/C-01
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2019-08

CONDITIONS: Patients Who Receive Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NPF-08 （1-day treatment） (Experimental)
  Interventions: Drug: NPF-08 （1-day treatment）
- NPF-08 （2-day split dose） (Experimental)
  Interventions: Drug: NPF-08 （2-day split dose）
- Moviprep（1-day treatment） (Active Comparator)
  Interventions: Drug: Moviprep（1-day treatment）

INTERVENTIONS:
Drug: NPF-08 （1-day treatment） — NPF-08 will be administered on the day of colonoscopy.
  Arms: NPF-08 （1-day treatment）
Drug: NPF-08 （2-day split dose） — NPF-08 will be administered at 2 days divided into the day before and on the day of colonoscopy.
  Arms: NPF-08 （2-day split dose）
Drug: Moviprep（1-day treatment） — Moviprep will be administered on the day of colonoscopy.
  Arms: Moviprep（1-day treatment）

SUMMARY:
To study non-inferiority of intestinal cleansing effect in both NPF-08 1-day treatment group and NPF-08 2-day split dose group to the cleansing effect in Moviprep® 1-day treatment group, for the subjects who will receive endoscopy large bowel. If the non-inferiority will be validated, superiority of intestinal cleansing effect in both groups of NPF-08 will be studied.

Furthermore, for the assessment of safety of NPF-08, the adverse events and adverse drug reactions observed after the administration to post-examination period will be studied, compared to those at Moviprep® 1-day treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese men and women aged 20 years or older at obtaining the written informed consent.
2. Patients who require colonoscopy (except for emergency colonoscopy)
3. Patients who have the ability to consent and submit the written informed consent by themselves.

Exclusion Criteria:

1. Patients who have or are suspected to have gastrointestinal obstruction.
2. Patients who have or are suspected to have intestinal perforation.
3. Patients who have or are suspected to have toxic megacolon.
4. Patients who have or are suspected to have gastric evacuation disorder (gastroparesis).
5. Patients with intestinal stenosis or high-grade constipation (stool frequency of 2 or less in a week or who have used laxative on a daily basis).
6. Patients with vomiting reflex or in whom accidental ingestion may occur.
7. Patients with a history of gastrointestinal surgery (except for appendicectomy).
8. Patients who were decided as glucose-6-phosphate dehydrogenase (G-6-PD) deficiency.
9. Patients with renal impairment (urea nitrogen: 25mg/dL or more, or creatinine: 2mg/dL or more)
10. Patients with hepatic dysfunction (total bilirubin: 3.0mg/dL or more, ALT: 100IU/L or more or AST: 100IU/L or more)
11. Patients who have undergone or require therapy due to high-grade cardiac disease (including angina pectoris or myocardial infarction)
12. Patients with high risk of arrhythmia (with a history or complications of QT prolongation, myocardial infarction, angina pectoris, cardiac failure or cardiomyopathy)
13. Patients with dehydration.
14. Patients who were diagnosed with active inflammatory bowel disease at screening period.
15. Inpatients due to the reasons other than endoscopy large bowel.
16. Patients who have undergone nutritional control using total parenteral nutrition or enteral nutrition.
17. Women who are or may be pregnant, lactating or wish to become pregnant during the trial period.
18. Patients with a history or high-risk of seizure.
19. Patients with a history of shock or hypersensitivity for the active ingredient of the investigational product.
20. Patients who have received the other investigational product within 4 months before the written informed consent or who are participating in the other clinical trials.
21. Patients in whom Investigator/Sub-Investigator decided not to be eligible for this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
The efficacy rate of overall intestinal cleansing effect evaluated by Endoscopic Image Evaluation Committee (EIEC). | 1day
  The bowel cleanliness at 5 colon segments (appendix/ascending colon, transverse colon, descending colon, sigmoid colon, rectum) will be evaluated. If the bowel cleanliness is "1" or "2" at all colon segments, it is judged as effective. Other cases will be judged as not effective.
  1. Almost no residue is found in the intestinal tract enabling good observation
  2. Residue remains but does not interfere the observation
  3. Residue interferes the observation
  4. A lot of residue makes unable to observe
  5. Unable to evaluate

SECONDARY OUTCOMES:
The efficacy rate of overall intestinal cleansing effect evaluated by colonoscopists | 1day
  The bowel cleanliness at 5 colon segments (appendix/ascending colon, transverse colon, descending colon, sigmoid colon, rectum) will be evaluated. If the bowel cleanliness is "1" or "2" at all colon segments, it is judged as effective. Other cases will be judged as not effective.
  1. Almost no residue is found in the intestinal tract enabling good observation
  2. Residue remains but does not interfere the observation
  3. Residue interferes the observation
  4. A lot of residue makes unable to observe
  5. Unable to evaluate
Colon cleansing effect by site | 1day
  The bowel cleanliness at 5 colon segments (appendix/ascending colon, transverse colon, descending colon, sigmoid colon, rectum) will be evaluated.
  1. Almost no residue is found in the intestinal tract enabling good observation
  2. Residue remains but does not interfere the observation
  3. Residue interferes the observation
  4. A lot of residue makes unable to observe
  5. Unable to evaluate
Evaluation based on Ottawa Bowel Preparation Scale | 1day
  Endoscopic operators will evaluate for colon cleansing degree at the bowel 5 sites (cecum/ascending colon, transverse colon, descending colon, sigmoid colon and rectum) based on the following 5 degrees (0-4) and the amount of fluid at overall bowel based on the following 3 degrees (0-2), and will also evaluate the status during operating normal endoscopy. Lower score indicates better cleansing effect.
Time from the initiation of dosing the investigational product to the completion of colon cleansing on the day of endoscopy. | 1day
  Clinical cooperator will determine the duration from the initiation of administration of the investigational product on the day of colonoscopy to the time when the cooperator will decide that colon cleansing will be completed as the discharged liquid will become transparent.
Dosage of the investigational product. | 1day or 2day
  Clinical cooperator will determine the dosage of the investigational product from the initiation of administration of the investigational product to the time when the cooperator will decide that colon cleansing will be completed as the discharged liquid will become transparent.
Concordance rate of intestinal cleansing effect between by EIEC members. | 1day
  For the evaluations of intestinal cleansing degree conducted at the primary endpoint, the concordance rate between by 3 members of EIEC will be investigated.
Concordance rate between the intestinal cleansing effect evaluated by EIEC and the endoscopic operators. | 1day
  For the evaluations of intestinal cleansing degree conducted at the primary endpoint and secondary endpoints, the concordance rate between the evaluations by EIEC and that by the endoscopic operators will be investigated.
Acceptability by subjects | 1day
  Subjects will evaluate the following points by selecting among 10 levels (circling the applicable figure): Taste of the investigational product; amount of the investigational product; amount of water you will drink after taking the investigational product; and acceptability of the pre-medication (will you choose the pre-medication at the next time?).

CONTACTS AND LOCATIONS:
Overall Officials: Hisatsugu Asada, Study Chair — Nihon Pharmaceutical Co., Ltd
Locations (13):
- Japan (13):
  - NPF-08 Trial Site 12, Abiko, Chiba
  - NPF-08 Trial Site 11, Kashiwa, Chiba
  - NPF-08 Trial Site 1, Maebashi, Gunnma
  - NPF-08 Trial Site 10, Kawasaki, Kanagawa
  - NPF-08 Trial Site 5, Yokohama, Kanagawa
  - NPF-08 Trial Site 9, Yokohama, Kanagawa
  - NPF-08 Trial Site 2, Chuo-Ku, Tokyo
  - NPF-08 Trial Site 3, Minato-Ku, Tokyo
  - NPF-08 Trial Site 4, Shinjuku-Ku, Tokyo
  - NPF-08 Trial Site 8, Hiroshima
  - NPF-08 Trial Site 13, Kouchi
  - NPF-08 Trial Site 6, Osaka
  - NPF-08 Trial Site 7, Osaka

REFERENCES:
- [Derived] Saito Y, Oka S, Tamai N, Kudo T, Kuniyoshi N, Shirakura T, Omae Y, Hamahata Y, Arai T, Tanaka S, Uedo N, Shimizu S, Fukuzawa M, Uraoka T, Ichinose S, Ogata H, Kobayashi K, Saito S, Tajiri H. Efficacy and safety of oral sulfate solution for bowel preparation in Japanese patients undergoing colonoscopy: Noninferiority-based, randomized, controlled study. Dig Endosc. 2021 Nov;33(7):1131-1138. doi: 10.1111/den.13930. Epub 2021 Mar 9. PMID 33476415